CLINICAL TRIAL: NCT02149797
Title: Prospective Randomized Comparative Study of New Single-incision Laparoscopic Cholecystectomy Technique, "Pick'n Roll", Versus Conventional Four-port Laparoscopic Cholecystectomy
Brief Title: Comparison of "Pick'n Roll" Single-incision Laparoscopic Cholecystectomy Technique, and Laparoscopic Cholecystectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsun Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Recep Aktimur, MD, Samsun Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SILC-PR vs. LC
Record Dates: First submitted 2014-05-21; First posted 2014-05-29 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Cholelithiasis
MeSH Terms: conditions — Cholelithiasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Four port laparoscopic cholecystectomy (Active Comparator): This group of patients undergone classical four port laparoscopic cholecystectomy
  Interventions: Procedure: Four port laparoscopic cholecystectomy
- SILC-Pick'n roll-Beginning (group I) (Active Comparator): This group of patients undergone single-incision laparoscopic cholecystectomy using our new technique called "Pick'n roll", this group was designed new intervention's beginning arm.
  Interventions: Procedure: SILC-Pick'n roll-Beginning (group I)
- SILC-Pick'n roll-Experienced (group II) (Active Comparator): This group of patients undergone single-incision laparoscopic cholecystectomy using our new technique called "Pick'n roll", this group was designed new intervention's experienced arm.
  Interventions: Procedure: SILC-Pick'n roll-Experienced (group II)

INTERVENTIONS:
Procedure: Four port laparoscopic cholecystectomy — Classical four port laparoscopic cholecystectomy
  Arms: Four port laparoscopic cholecystectomy
Procedure: SILC-Pick'n roll-Beginning (group I) — SILC-PR was performed by the intraumbilical single port technique. A 10-mm, 30º scope was used. The surgeon was elevated gallbladder fundus with left hand using grasper in whole operation. If required, infindibulum was freed with monopolar hook. A 2.0 straight needle was inserted through the right of the falciform ligament, grasped with a laparoscopic needleholder using by surgeon's right hand, and passed through the Hartmann's pouch at the lowest point. To allow free manipulation, the passing suture with needle was turned around the suture to form a "half-knot". The needle was passed back out from the right of the midclavicular line. An assistant was grasped two ends of the suture and with the help of right or left hand dominant pulling tension, critical view of safety was provided
  Arms: SILC-Pick'n roll-Beginning (group I)
Procedure: SILC-Pick'n roll-Experienced (group II) — Similar technique of SILC-Pick'n roll-Beginning (group I) was used
  Arms: SILC-Pick'n roll-Experienced (group II)

SUMMARY:
Cholecystectomy is one of the most common operation performed by general surgeons. Since, first video-laparoscopic cholecystectomy in 1987, laparoscopic cholecystectomy (LC) has become the gold standard treatment for benign biliary disease. In daily practice, LC has increased general surgeons familiarity to video-laparoscopic operations and has become the first step to search more minimally invasive techniques and to perform advanced laparoscopic operations. In order to move forward the minimal invasive surgery concept with less surgical trauma and better cosmetic results, surgeons firstly reduced the number of incision and ports, then the idea of totally eliminating skin incisions through the use of natural orifices was implemented in selected cases.

In theory, minimal incision must provide minimal postoperative pain and better cosmetic results. With the use of single-incision laparoscopic cholecystectomy (SILC), this purpose is achieved by means of cosmesis but providing minimal postoperative pain is still controversial. Recent reports on, LC vs. SILC showed significantly favorable cosmetic benefit, comparable complication rate and hospital stay with SILC, but the mean operation time was significantly longer. Today, lack of standardized operation technique, the need for specialized instruments, the fear of inability to apply safe cholecystectomy principles, longer operation time, cost-effectivity and advanced laparoscopic experience are still limiting factor to performing SILC.

The aim of this prospective randomized controlled trial is to compare gold standard LC and SILC using our new technique called "Pick'n roll" (SILC-PR). Our goal was to provide critical view of safety and safe cholecystectomy principles on SILC, improve operator ergonomics and shorten operation time while eliminating the need for specialized instruments.

DETAILED DESCRIPTION:
A pilot study was conducted, with ten patients who were planned to perform laparoscopic cholecystectomy after approval by the ethics committee of Ondokuz Mayis University, Samsun, Turkey. Among ten patients, five patients were undergone LC, and another five were undergone SILC-PR.

The sample size was calculated from the pilot study. Simple consecutive allocation method was used to randomly divide the subjects into LC (classical four port technique), and SILC-"Pick'n roll" (PR) beginning and experienced groups. Each group contained 20 patients. The randomization was achieved regardless of demographic characteristics, by Dr. N. O.

One surgeon was performed all operation (Dr. R. A.). Patient's data were recorded by Dr. K. Y. At the end of the study, the data were analysed by Dr. S. C. and Dr. E. C. in a blinded manner to avoid bias

Surgical Procedures The technique used for LC was the conventional four-trocar approach (10-mm optic at the umbilicus, 10-mm trocar in the epigastrium and two 5-mm trocars in the right upper abdomen).

For SILC-PR, the patient was positioned supine on the operating table, once the access is gained into the abdomen, the patient re-positioned to reverse trendelenburg and left tilt. The surgeon stands on the left side of the patient and the assistant stands opposite him during the placement of the single-port device. SILC-PR was performed by the single-incision, single port technique using The OCTOTMPort (Dalimsurg, Seoul, Korea). The OCTOTMPort is a re-usable single-port device that contains two 5-mm, one 10-mm and one 12-mm port through the same port. Surgical access to the abdomen was obtained through an intraumbilical 2.5 cm incision from 12 o'clock to 6 o'clock. The OCTOTMPort was inserted and pneumoperitoneum was created up to an abdominal pressure of 15 mmHg. A 10-mm, 30º traditional scope (Karl Storz, Tuttlingen, Germany) was inserted through inferior placed 10-mm port, by the assistant who positioned on the patient's left side, and the peritoneal cavity was examined. If the stomach was distended, a nasogastric tube insertion was requested from the anesthesiologist. The surgeon introduced an Endo Grasp™ (Covidien, Mansfield, MA, USA) with left hand and elevated gallbladder fundus to assess the mobility of the gallbladder infindibulum, constant fundus retraction was used in whole operation by this instrument. In the presence of omental attachments, the gallbladder infindibulum was freed with monopolar hook device which holding by the surgeon's right hand, under the traction of the fundus. Once the gallbladder infindibulum freed from the attachments or clearly seen in first examination next step of the operation was launched. A 2.0 multifilament straight atraumatic needle was inserted through the surgeon's left of the falciform ligament with simultaneous palpation of the abdominal wall for optimum insertion site. The needle was grasped with a laparoscopic needleholder using by surgeon's right hand, and the needle was passed through the Hartmann's pouch at the lowest accessible point. To allow infindibulum retraction, wide triangulation and free Hartmann's pouch manipulation like "puppeteer movement", the passing suture with needle was turned around the afferent suture and a "half-knot" was created. The needle was passed back of the abdomen from the surgeon's left of the midclavicular line, with simultaneous palpation of the abdominal wall for optimum site. After this point, an assistant or a nurse was grasped two ends of the suspensory suture with clamps. With the help of fundus retraction and assistant's right or left hand dominant pulling tension on the suture, classical Hartmann's pouch retraction similar to LC technique was provided. Dissection of Calot's triangle and removal of gallbladder from the liver bed are possible in almost all cases with the use of aforementioned "Pick'n roll technique" and a hook diathermy.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic cholelithiasis

Exclusion Criteria:

* Acute cholecystitis (diagnosed on ultrasound or elevated inflammatory serum markers)
* Choledocholithiasis
* Less than 18 years old
* American Society of Anesthesiologist (ASA) grade IV or V.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Operation time | Up to 1.5 hours

SECONDARY OUTCOMES:
Conversion to open or classical laparoscopic cholecystectomy | Up to 1.5 hours
Insertion of additional port/ports. | Up to 1.5 hours
Intraoperative complication | Up to 1.5 hours
Lenght of hospital stay | Up to 3 days
Postoperative complication rate | Up to 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Recep Aktimur, Principal Investigator — Samsun Education and Research Hospital, Samsun, Turkey
Locations (1):
- Samsun Education and Research Hospital, Department of General Surgery, Samsun, Turkey, Samsun, Turkey (Türkiye)

REFERENCES:
- [Background] Sajid MS, Ladwa N, Kalra L, Hutson KK, Singh KK, Sayegh M. Single-incision laparoscopic cholecystectomy versus conventional laparoscopic cholecystectomy: meta-analysis and systematic review of randomized controlled trials. World J Surg. 2012 Nov;36(11):2644-53. doi: 10.1007/s00268-012-1719-5. PMID 22855214
- [Background] Philipp SR, Miedema BW, Thaler K. Single-incision laparoscopic cholecystectomy using conventional instruments: early experience in comparison with the gold standard. J Am Coll Surg. 2009 Nov;209(5):632-7. doi: 10.1016/j.jamcollsurg.2009.07.020. Epub 2009 Sep 11. PMID 19854405
- [Background] Lai EC, Yang GP, Tang CN, Yih PC, Chan OC, Li MK. Prospective randomized comparative study of single incision laparoscopic cholecystectomy versus conventional four-port laparoscopic cholecystectomy. Am J Surg. 2011 Sep;202(3):254-8. doi: 10.1016/j.amjsurg.2010.12.009. PMID 21871979